CLINICAL TRIAL: NCT02361359
Title: Preoperative Catastrophizing Predicts Pain Outcome After Shoulder, Knee and Hip Arthroplasty
Status: Completed | Type: Observational
Sponsor: Hospital Ambroise Paré Paris (Other)
Responsible Party: Principal Investigator, Shahnaz Klouche, MD, Physician responsible of clinical research, Hospital Ambroise Paré Paris
Other Study IDs: APR012014
Record Dates: First submitted 2015-02-06; First posted 2015-02-11 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Osteoarthritis; Chronic Pain; Catastrophization
Keywords: Arthroplasty
MeSH Terms: conditions — Osteoarthritis; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Psychological questionnaires

SUMMARY:
Psychologic status is associated with poor outcome after joint arthroplasty and perhaps chronic pain. To enhance the therapeutic effect of a psychologic intervention, the specific disorders or pain-related beliefs that contributed to chronic pain should be identified. We therefore determined whether specific psychologic disorders (depression, anxiety disorder) or health-related beliefs (self-efficacy, pain catastrophizing) are associated with chronic pain after joint arthroplasty for osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* joint arthgroplasty (shoulder, hip ou knee)
* osteoarthritis

Exclusion Criteria:

* previous surgery in the same joint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergo joint arthroplasty (shoulder, hip ou knee) for osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-01; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Pain score | 1 year postoperatively

SECONDARY OUTCOMES:
Functional score | 1 year postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Ambroise Paré Paris, Boulogne-Billancourt, France

REFERENCES:
- [Derived] Hardy A, Sandiford MH, Menigaux C, Bauer T, Klouche S, Hardy P. Pain catastrophizing and pre-operative psychological state are predictive of chronic pain after joint arthroplasty of the hip, knee or shoulder: results of a prospective, comparative study at one year follow-up. Int Orthop. 2022 Nov;46(11):2461-2469. doi: 10.1007/s00264-022-05542-7. Epub 2022 Aug 23. PMID 35999466